CLINICAL TRIAL: NCT05827250
Title: Passive Infrasound-to-ultrasound Vibrome Biosignatures of Lung Development in Newborn Infants
Brief Title: Vibroacoustic Study of Lung Development in Newborn Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Level 42 AI, Inc. (Industry)
Collaborators: Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: L42CVP-0007
Record Dates: First submitted 2023-03-18; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Prematurity; Premature Birth; Premature Lungs; Prematurity; Extreme
Keywords: infrasound; vibrome; vibroacoustics
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonatal Profile: LUSS will be obtained twice a week on the following schedule for the duration of each subject's NICU stay.
  Day of life (DOL): 7+/-1, 10+/-1, and 14+/-1 Depending on length of stay, within +/-2 days of: DOL 17, 21, 24, 28, 31, 35, 38, 41, 44, 48, 51, 56, and 60.
  Interventions: Device: imPulse Tor

INTERVENTIONS:
Device: imPulse Tor — The imPulse-Tor system passively collects audible sounds and inaudible vibrations spanning the infrasound-to-ultrasound frequency range, as well as cardiac electrical signals. The device can be safely placed directly on the chest wall to obtain readings.
  imPulse System vibroacoustic recording (VAR) will be performed twice daily till discharge. An attempt will be made to have at least a 6+/-2 hr gap between the two recordings.
  Other Names: imPulse Tor infrasound-to-ultrasound e-stethoscope plus multi-lead ECG

SUMMARY:
Investigators hypothesize that premature newborns with poor cardiopulmonary performance have higher morbidities and poorer physical and cognitive developmental outcomes.

Investigators further hypothesize that audible sounds combined with novel inaudible vibrations above and below human perception interpreted with transparent and auditable AI algorithms can detect and identify early gas and fluid movement anomalies not uncovered by conventional tools in an non-invasive, easy, fast, and low cost examination.

DETAILED DESCRIPTION:
Worldwide preterm birth (<37 weeks of gestation) affects approximately 10% of live births and is the leading cause of death in children less than 5 years of age. Preterm birth disrupts normal lung development leading to several respiratory complications in the neonatal period and later in life. Consequently, factors that negatively affect prenatal and early life respiratory growth can compromise the achievement of "personal-best lung function".

This novel study will generate normative, audible/inaudible frequencies, visible/invisible frequencies, and perceptible/imperceptible energies, termed vibrome biosignatures, of cardiopulmonary development and function during early postnatal development. Once baseline patterns are established, future studies will be designed to characterize vibrome biosignature differences across acute neonatal respiratory problems, such as respiratory distress syndrome, meconium aspiration, sepsis, persistent pulmonary hypertension, and congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants include all infants admitted to the NICU.

Exclusion Criteria:

* There are no exclusions to enrollment in this study.

Ages: 0 Years to 2 Years | Sex: All
Age Groups: Child
Study Population: All infants admitted to the NICU
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-09-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Gestational age change in lung vibroacoustics | through study completion, an average of 6 weeks
  Correlate the relationship of vibroacoustic measurements (i.e., vibroacoustic wave's maximum pressure fluctuations, represented by the base unit known as a Pascal) with gestational age (wks) as modified by clinical status.

CONTACTS AND LOCATIONS:
Overall Officials: Pinaki Panigrahi, MD, PhD, Principal Investigator — Georgetown University Medical Center Pediatrics
Locations (1):
- Medstar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing language not included in consent for this pilot study